CLINICAL TRIAL: NCT02977182
Title: The Effect of Lymphedema Treatment for the Management of Blunt Facial Trauma
Brief Title: Lymphedema Treatment for Blunt Facial Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Responsible Party: Principal Investigator, Danielle Tatum, Academic Research Director, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9521
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Post-traumatic Facial Edema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): The control group will receive standard speech therapy treatments but not lymphedema treatment and will serve as the baseline for comparison for assessment of the effects of CDT.
- Active Treatment Group (Experimental): The active treatment group will receive standard speech therapy treatments in addition to complete decongestive therapy from a certified Speech Language Pathologist (CCC-SLP) trained in CDT.
  Interventions: Other: Complete Decongestive Therapy (CDT)

INTERVENTIONS:
Other: Complete Decongestive Therapy (CDT) — CDT is a multimodal therapy consisting of four components: manual lymph drainage, compression wrapping, exercise, and skin care
  Arms: Active Treatment Group

SUMMARY:
Injuries to the face caused by traumatic events such as motor vehicle collisions, assault, and falls can result in facial trauma, which can result in swelling and disfiguration that impairs the important functions of the face, sometimes to a life threatening degree. These injures and the resultant swelling can also precipitate psychological and social consequences.

Lymphedema is an abnormal amount of fluid that causes swelling, usually in the arms or legs. The most common presentation of lymphedema is in the upper extremities due to breast cancer treatment (Maclellean RA et al). As such, standards of care for management of lymphedema are primarily derived from the cancer research literature and involve the extremities (Moffatt CJ. 2003 QJM). The current gold standard treatment for patients with extremity lymphedema is complete decongestive therapy (CDT) (Zuther 2013). CDT is a multimodal therapy consisting of four components: manual lymph drainage, compression wrapping, exercise, and skin care (Zuther 2013).These same therapeutic techniques of CDT have been employed at Our Lady of the Lake Regional Medical Center (OLOLRMC) and adapted to treat patients with facial trauma with anecdotally good results primarily related to cosmesis. To the best of our knowledge, no clinical studies examining the effect of lymphedema treatment in the management of blunt facial trauma currently exist.. Beyond the consideration of cosmesis, we also seek to determine if this intervention improves clinical outcomes such as time to swallowing and reduced time utilizing mechanical ventilation. This study will prospectively evaluate the use of complete decongestive therapy to test the hypothesis that this intervention results in improved clinical outcomes in patients with blunt facial trauma.

DETAILED DESCRIPTION:
Introduction The face is an anatomically complex structure, consisting of skin, muscles for both fine and gross motor functions, a complex bony structure, and vital sensory organs. These structures allow one to eat, breathe, see, hear, and speak. Injuries to the face caused by traumatic events such as motor vehicle collisions, assault, and falls can result in facial trauma, which can result in swelling and disfiguration that impairs the important functions of the face, sometimes to a life threatening degree. These injures and the resultant swelling can also precipitate psychological and social consequences.1-3 Lymphedema is an abnormal amount of fluid that causes swelling, usually in the arms or legs. Though lymphedema can occur as a result of trauma, it is most commonly associated with side effects of certain cancer-related treatments such as radiation therapy and lymph node removal. The most common presentation of lymphedema is in the upper extremities due to breast cancer treatment.4 As such, standards of care for management of lymphedema are primarily derived from the cancer research literature and involve the extremities.5 The current gold standard treatment for patients with extremity lymphedema is complete decongestive therapy (CDT).6 CDT is a multimodal therapy consisting of four components: manual lymph drainage, compression wrapping, exercise, and skin care.6 Manual lymph drainage (MLD) is a delicate form of massage designed to improve tissue and cellular health by facilitating fluid removal from edematous areas. Compression wrapping utilizes compression garments or short stretch compression bandages and is primarily used in the acute (or intensive) phase of CDT as a means to reinstate sufficient resistance to skin tissues whose elastic fibers are damaged by lymphedema. Exercise, especially when combined with compression, improves removal of fluid from the affected area. Finally, skin care treatments keep skin clean and moisturized to reduce infections that can occur with lymphedema.6 These same therapeutic techniques of CDT have been employed at Our Lady of the Lake Regional Medical Center (OLOLRMC) and adapted to treat facial edema in patients with facial trauma with anecdotally good results in terms of cosmesis. To the best of our knowledge, no clinical studies examining the effect of lymphedema treatment in the management of blunt facial trauma currently exist. Beyond the consideration of cosmesis, we also seek to determine if this intervention improves clinical outcomes such as time to swallowing and reduced time utilizing mechanical ventilation. This study will prospectively evaluate the use of complete decongestive therapy to test the hypothesis that this intervention results in improved clinical outcomes in patients with blunt facial trauma.

Specific Aims Specific Aim I: To determine whether complete decongestive therapy can significantly reduce facial lymphedema as measured by a previously established facial composite scoring protocol.

Specific Aim II: To determine whether complete decongestive therapy can improve clinical outcomes for patients with facial trauma Study Objective and Endpoints Study Objective The primary objective of this study is to determine the effect(s), if any, of complete decongestive therapy in the management of facial trauma.

Primary Endpoint The primary endpoint will be the composite facial score measured on the day of discharge from the Trauma Neuro Critical Care (TNCC) intensive care unit (ICU) at OLOLRMC. This measurement is based on the Head & Neck Lymphedema (HNL) program at MD Anderson Cancer Center (MDACC) whose standard evaluation protocol includes specific point-to-point measurements of the face (Smith & Lewin 2010; Smith and Lewin 2014). A series of key facial measurements are totaled to provide a "composite facial score". Based on the clinical experience at MDACC with more than 150 patients, their HNL program has developed criteria to define clinically detectable improvements in external HNL. Those criteria are a drop in lymphedema stage or a minimum threshold of 2% reduction in the composite measurement equating to at least a 2-cm change in absolute values (Smith & Lewin 2014).

Secondary endpoints

Because the facial and neck composite scores only provide evaluation of the extent of edema, we also seek to assess patient outcomes with regards to the following:

1. Stage of lymphedema as defined by the MDACC HNL edema rating scale
2. Number of mechanical ventilation days
3. Narcotic pain medicine utilization
4. Steroid utilization
5. Pain scale scores as determined by the Visual Analog Scale or the adult non-verbal pain score
6. Time to swallowing
7. ICU length of stay (ICULOS)
8. Hospital length of stay (LOS)

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients 18 years of age or older
* Presence of facial trauma as determined by X-ray or computed tomography (CT)
* Presence of face/neck lymphedema characterized as at least Stage 1 on the MD Anderson Cancer Center's Head and Neck Lymphedema (HNL) rating scale

Exclusion Criteria:

* Less than 18 years of age

  * Presence of injury to the carotid artery or jugular veins
  * Presence of upper quadrant deep vein thrombosis
  * Presence of known infection
  * Unwilling or unable to consent (or unable to find an appropriate surrogate)
  * Pregnant
  * Expected death within 24 hours of enrollment, or desire by patient of family to pursue palliative rather than aggressive, supportive care
  * Inability to speak English such that assessment of primary endpoints would not be feasible
  * Prisoners
  * Patients previously enrolled in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Composite facial score | Up to 2 weeks
  This measurement is based on the Head & Neck Lymphedema program at MD Anderson Cancer Center whose standard evaluation protocol includes specific point-to-point measurements of the face which are totaled to provide a composite facial score.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Tatum, PhD, Study Director — OUR LADY OF THE LAKE RMC
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glynn SM, Asarnow JR, Asarnow R, Shetty V, Elliot-Brown K, Black E, Belin TR. The development of acute post-traumatic stress disorder after orofacial injury: a prospective study in a large urban hospital. J Oral Maxillofac Surg. 2003 Jul;61(7):785-92. doi: 10.1016/s0278-2391(03)00239-8. PMID 12856251
- [Background] Rankin M, Borah GL. Perceived functional impact of abnormal facial appearance. Plast Reconstr Surg. 2003 Jun;111(7):2140-6; discussion 2147-8. doi: 10.1097/01.PRS.0000060105.63335.0C. PMID 12794453
- [Background] Maclellan RA, Couto RA, Sullivan JE, Grant FD, Slavin SA, Greene AK. Management of Primary and Secondary Lymphedema: Analysis of 225 Referrals to a Center. Ann Plast Surg. 2015 Aug;75(2):197-200. doi: 10.1097/SAP.0000000000000022. PMID 24691335
- [Background] Glynn SM, Shetty V, Elliot-Brown K, Leathers R, Belin TR, Wang J. Chronic posttraumatic stress disorder after facial injury: a 1-year prospective cohort study. J Trauma. 2007 Feb;62(2):410-8; discussion 418. doi: 10.1097/01.ta.0000231556.05899.b0. PMID 17297333
- [Background] Moffatt CJ, Franks PJ, Doherty DC, Williams AF, Badger C, Jeffs E, Bosanquet N, Mortimer PS. Lymphoedema: an underestimated health problem. QJM. 2003 Oct;96(10):731-8. doi: 10.1093/qjmed/hcg126. PMID 14500859
- [Background] Cohen MD. Complete decongestive physical therapy in a patient with secondary lymphedema due to orthopedic trauma and surgery of the lower extremity. Phys Ther. 2011 Nov;91(11):1618-26. doi: 10.2522/ptj.20100101. Epub 2011 Aug 25. PMID 21868611